CLINICAL TRIAL: NCT01379196
Title: Use of Azithromycin as Immunomodulatory Therapy in Grave&Apos;s Orbitopathy
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Patients were not interested in enrolling
Sponsor: Rabin Medical Center (Other)
Responsible Party: Principal Investigator, kalish hadas, Chief, Neuro-Ophthalmology Unit, Rabin Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0427-10-RMC
Record Dates: First submitted 2011-05-11; First posted 2011-06-23 (Estimated); Last update posted 2017-04-27 (Actual); Status verified 2017-04

CONDITIONS: Graves Ophthalmopathy
Keywords: Graves Orbitopathy; Macrolide antibiotics; Inflammation; Clinical Activity Score
MeSH Terms: conditions — Graves Ophthalmopathy; Inflammation | interventions — Azithromycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Azithromycin PO three times weekly (Experimental): Tablets Azithromycin 500 mg PO three times weekly for three months
  Interventions: Drug: Azithromycin

INTERVENTIONS:
Drug: Azithromycin — Tab. Azithromycin 500 mg PO three times weekly for 3 months
  Other Names: AZITRO

SUMMARY:
The purpose of this study is to examine the effects of Azithromycin (a macrolide class antibiotic), given three times weekly, for patients with active moderate-severe, non sight-threatening, Graves Orbitopathy.

Indices for follow-up will include:

* Clinical activity score
* Anti-TSH receptor antibody levels
* Thickening of extraocular muscles per ultrasound
* Quality of life score for Graves Orbitopathy patients

DETAILED DESCRIPTION:
Graves Orbitopathy (GO) is an autoimmune inflammatory disorder causing visual morbidity, cosmetic morbidity and interference with quality of life. The disease has an inflammatory stage and a non-inflammatory, fibrotic stage.

Treatment of inflammatory stage moderate-severe GO includes steroids, as recommended by the EUGOGO consortium. However, the length of treatment needed and the risk of steroid side-effects may lead to multiple undesired treatment induced morbidity.

Antibiotics of the macrolide group posses known immune-modulatory effects that are separate from their antibacterial mode of action. This mode of action has lead to the routine use of macrolide antibiotics for delaying graft rejection following lung transplants.

We propose to test the effect of this class of antibiotics for non-sight threatening, moderate-severe, inflammatory GO.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Graves Orbitopathy
* Clinical activity score higher than 2
* Must be able to swallow tablets

Exclusion Criteria:

* sight-threatening Graves Orbitopathy
* Diplopia in primary gaze
* Macrolide allergy or intolerance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-05; Primary Completion 2014-11 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Change in clinical activity score between baseline and after three months | Three months
  Change in the clinical activity score between baseline and after 3 months
  (Clinical Activity Score is a validated index of Graves Ophthalmopathy that assigns one point to the presence of: 1.spontaneous retrobulbar pain, 2. pain on up/downgaze, 3. redness of eyelids, 4. redness of conjunctiva, 5. swelling of eyelids, 6. inflammation of caruncle/plica, 7. chemosis). The maximal clinical activity score is thus 7.

SECONDARY OUTCOMES:
Measurement of extraocular muscle thickening | 3 months
  Ultrasonic measurement of extraocular muscle thickening
ANTI TSH Receptor antibody levels | 0, 3 and 6 months
  Serum measurements of ANTI TSH Receptor antibody levels

CONTACTS AND LOCATIONS:
Overall Officials: Hadas Kalish, MD, Principal Investigator — Neuro-Ophthalmology Unit, Rabin Medical Center, Petah Tikva 49100 Israel

IPD SHARING:
Plan to Share IPD: Undecided